CLINICAL TRIAL: NCT04471506
Title: High-intensity Interval Training and Mindfulness Breathing Induce Hormonal and Metabolic Effects and Alter Tumor Marker Levels in Obese Postmenopausal Women: A Randomized Controlled Trial
Brief Title: Effect of Interval Aerobic Training and Mindfulness Breathing on Hormonal, Metabolic, and Tumor Markers in Postmenopausal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P.T.REC/012/004118
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group will receive interval training and mindfulness breathing (Other): exercise program in form of a cycling protocol which will be comprised 5 minutes of warming up before exercise initiation and another 5 minutes for cooling down by the end of the exercise session in the form of slow pedaling (50% of PHR). The work interval also will be consisted of 8-12 cycling intervals (60s cycling work interval with 120s of passive rest or low-intensity cycling (70% of PHR) between work intervals that progressively will be reduced until reaching 90s by the end of the exercise program). Mindful breathing is a exercise that involves using breathing as an object of attention. 15-minute mindful breathing intervention will be adapted. It consists of the following three steps: (a) adopt a physical posture, (b) establish a mindfulness anchor, and (c) maintain mindfulness
  Interventions: Other: interval training; Other: diet recommendations; Other: mindfulness breathing
- diet recommendations (Other): The control group will receive diet recommendations. The volunteers will follow diet recommendations for 12 weeks
  Interventions: Other: diet recommendations

INTERVENTIONS:
Other: interval training — Ixercise program in form of a cycling protocol which will be comprised 5 minutes of warming up before exercise initiation and another 5 minutes for cooling down by the end of the exercise session in the form of slow pedaling (50% of PHR). The work interval also will be consisted of 8-12 cycling intervals (60s cycling work interval with 120s of passive rest or low-intensity cycling (70% of PHR) between work intervals that progressively will be reduced until reaching 90s by the end of the exercise program).
  Arms: study group will receive interval training and mindfulness breathing
Other: diet recommendations — the control group will follow diet recommendations for 12 weeks
Other: mindfulness breathing — Mindful breathing is a exercise that involves using breathing as an object of attention. 15-minute mindful breathing intervention will be adapted. It consists of the following three steps: (a) adopt a physical posture, (b) establish a mindfulness anchor, and (c) maintain mindfulness
  Arms: study group will receive interval training and mindfulness breathing

SUMMARY:
PURPOSE:

to determine the effect of interval training and mindfulness breathing on sex hormones, metabolic and tumor markers

BACKGROUND:

Cancer is one of death top causes in many countries1. In Egypt for example, cancer incidence is 157.0 per 100 000 women with probability increasing up to three-fold by 2050 especially in older adult women2. Who exhibit multiple factors leading to cancer including but not limited to physical inactivity and postmenopausal obesity which considered the starting point of developing insulin resistance3.

High blood insulin level stimulates cancer progression by enhancing cell proliferation, decreasing cells apoptosis, increased level of fatty acids in conjunction with higher tumor cell formation capacity invasion and survival4. Moreover, high level of insulin resistance and adipose tissue increase the hormonal level of estradiol and testosterone coupled with lower SHBG level.

It was noticed that being postmenopausal women with high adipose tissue content will increase the risk of having cancer in which adipose tissue is considered as the main source of steroids hormones that functioning in a different way rather than in premenopausal age. Based on the mentioned underlying conditions, postmenopausal women subjected to have variable types of cancer such as breast, endometrial, stomach, etc6.

So, regular screening of cancer incidence especially in high-risk women through tumor indicators is necessitated to work against further cancer progression. CEA and CA125 are low-cost tumor blood biomarkers used widely for early cancer identification, recurrence monitoring and follow up which linked to proinflammatory cytokines production

.

HYPOTHESES:

may have no effect to interval training and mindfulness breathing on sex hormones , metabolic and tumor markers in postmenopausal women

RESEARCH QUESTION:

Is there effect to interval training and mindfulness on sex hormones , metabolic and tumor markers in postmenopausal women?

DETAILED DESCRIPTION:
HIIT group involved in an exercise program three times per week for three months in form of cycling protocol which will comprise 5 minutes warming up before exercise initiation and another 5 minutes for cooling down by the end of exercise session in form slow pedaling (50% of PHR). The work interval also will comprise 8-12 cycling intervals (60s cycling work interval with 120s of passive rest or low-intensity cycling (70% of PHR) between work intervals that progressively will be reduced until reaching 90s by the end of the exercise program)17. Each work interval will be maintained at a range of 50-70 rpm (cycle revolutions) with a speed between 20 and 40 km/h. Exercise intensity will be ≥ 85% of peak heart rate (PHR) according to the Karvonen formula18.

which corresponds to 8-10 points on the modified Borg scale19. The exercise will be supervised along the first week only with guidance to ensure that each participant masters the optimal exercise procedure.

The participants will be equipped with a pulse oximeter for continuous monitoring of the heart rate prior to the start, during or just after the completion of the exercise session .Also, Mindful breathing is a exercise that involves using breathing as an object of attention. 15-minute mindful breathing intervention will be adapted. It consists of the following three steps: (a) adopt a physical posture, (b) establish a mindfulness anchor, and (c) maintain mindfulness . Healthy diet instructions will be recommended for those non-dietitian obese women without following specific diet programs that could influence our results.

ELIGIBILITY:
Inclusion Criteria:

* Sixty Postmenopausal women (55-65 y)
* Body mass index (BMI) ranged from 35 to 39.9 kg/m2
* Postmenopausal more than 2 years

Exclusion Criteria:

* • women receiving weight-reduction interventions

  * taking lipid lowering drugs
  * regular medications(e.g., β-blockers, α-blockers, digoxin, diuretics, aspirin, nitrates, Presently using sex hormones)
  * having active chronic illness (e.g., rheumatoid arthritis, hyperthyroidism, and inflammatory bowel disease) and diabetes mellitus or other (unstable) endocrine-related diseases
  * cognitive impairment that will make it difficult to partake in the study
  * presence of malignant disease
  * blood donation within the last 30 days
  * Participation as a subject in any type of study or research during the prior 90 days
  * smoking

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
insulin resistance | 12 weeks
  insulin resistance will be measured by homeostasis model assessment (HOMA) index of change of insulin-resistance by homeostasis model assessment insulin resistance ( HOMA -IR )index
sex hormones | 12 weeks
  change of sex hormones level (e.g. estradiol ,testosterone. sex hormone binding globin )'
blood lipids | 12 weeks
  blood lipids will be measured by blood analysis,
tumor markers | 12 weeks
  tumor markers will be measured by blood analysis,

CONTACTS AND LOCATIONS:
Overall Officials: marwa m elsayed, phd, Principal Investigator — lecturer at physical therapy faculty cairo university
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: one year after completion the study
Access Criteria: students and scientific researchers will be allowed to access
URL: http://Scholar.cu.edu.eg/p_t